CLINICAL TRIAL: NCT00340392
Title: Isolation and Characterization of Mammary Stem Cells
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906140; 06-C-N140; NCT00900315 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-03-23

CONDITIONS: Stem Cells
Keywords: Mammary Stem Cells; Breast Cancer; Cancer Stem Cells; Gene Expression Profiling
MeSH Terms: conditions — Breast Neoplasms

SUMMARY:
Background:

* Cancer stem cells in breast cancer have been identified as a small population of tumor cells whose self-renewal mechanism is highly deregulated. This deregulation seems to be necessary for cancer to develop.
* These cells can be identified by certain surface markers that overlap with markers associated with normal embryonic stem cells.

Objective: To isolate tumor stem cells using the same methods generally used to isolate human embryonic stem cells.

Eligibility:

* Tissue samples will be obtained from the human cooperative network.
* Samples will include normal tissues from individuals who have no opportunistic diseases and from individuals with cancer.

Design: Breast cancer stem cells will be isolated, grown in the laboratory and characterized.

DETAILED DESCRIPTION:
Cancers are composed of heterogeneous populations of cells with varying degrees of proliferative capacity and ability to reconstitute tumors when transplanted into nude or SCID mice.

Recently, cancer stem cells have been identified as a small population of tumor cells which possess the stem cell properties in that their self-renewal pathway is highly deregulated. This deregulation seems to be the prerequisite for the development of cancer.

ELIGIBILITY:
* INCLUSION CRITERIA:

The tissue samples will come from the human cooperative network. They have their own set of criteria. We are requesting tissue samples from individuals that are normal as well as those who have cancer.

EXCLUSION CRITERIA:

The tissue samples will come from the human cooperative tissue network and we are asking for normal samples from individuals who don't have any opportunistic diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-04-07; Study Completion 2011-03-23

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States